CLINICAL TRIAL: NCT01862068
Title: Neutrophils Function and Identification of Prognostic Factors in Granulomatosis With Polyangiitis (Formerly Named Wegener's Granulomatosis).
Brief Title: Neutrophils as Prognostic Factors in Granulomatosis With Polyangiitis (Formerly Named Wegener's Granulomatosis)
Acronym: NeutroVasc
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI 10017
Record Dates: First submitted 2013-01-01; First posted 2013-05-24 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Granulomatosis With Polyangiitis
Keywords: Pronostic factors; Neutrophils; Granulomatosis with polyangiitis; Microscopic polyangiitis; ANCA associated vasculitis; Proteomics
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- GPA patients: GPA patients with an active disease at inclusion
  Interventions: Other: Blood samples and clinical data
- MPA patients
  Interventions: Other: Blood samples and clinical data
- Healthy Blood Donors
  Interventions: Other: Blood sample
- Atherosclerotic patients
  Interventions: Other: Blood samples and clinical data
- EGPA (Eosinophilic Granulomatosis With Polyangiitis)
  Interventions: Other: Blood samples and clinical data

INTERVENTIONS:
Other: Blood samples and clinical data — Blood samples will be performed at inclusion and at 12 months from all patients (4 groups GPA, MPA, EGPA and Atherosclerotic patients)
  Groups: Atherosclerotic patients; EGPA (Eosinophilic Granulomatosis With Polyangiitis); GPA patients; MPA patients
Other: Blood sample — Blood sample will be performed at inclusion from all healthy patients
  Groups: Healthy Blood Donors

SUMMARY:
Anti-neutrophil cytoplasm antibodies (ANCA)-associated vasculitis are rare diseases characterized by inflammation of blood vessels. Among the numerous cell types that play a role in vasculitis, one of the key actors is the neutrophil. Neutrophils are equipped with very powerful molecules that they use to destroy the invading microbes. Therefore, the mechanisms controlling neutrophil activation should be tightly controlled. If that is not the case, neutrophils may destroy the tissues of the host. This is what happens during chronic inflammation in vasculitis. Autoantibodies directed against neutrophils, ANCA, produced thus demonstrating that neutrophils are also targets of the immune system in these diseases. In addition, molecular studies provided evidence that genes normally silenced in mature neutrophils under normal conditions can be re-expressed in neutrophils from patients with ANCA-associated vasculitis thus strongly suggesting a profound deregulation of neutrophil functions in these conditions. Notably, the investigators have preliminary data showing that neutrophils from patients with granulomatosis with polyangiitis (GPA, formerly Wegener's granulomatosis), an ANCA-associated vasculitis, interfere with the normal phase of resolution of inflammation.

The objective of the investigators' study is to understand the mechanisms underlying this increased activation state and determine if neutrophils could be used to define prognostic markers by clinicians to optimize patients' care. Therefore, the investigators plan to study the expression of proteins implicated in GPA pathophysiology at the membrane of neutrophils when they undergo apoptosis. The investigators will also study the deregulation of protein expression in neutrophils. This point will be the molecular translation of neutrophil deregulation. This technique is powerful and well adapted to identify by mass spectrometry the proteins that will be differentially expressed between the control and the disease state. After identification of proteins differentially expressed in patients with GPA, the investigators will further investigate whether their expression is modulated during the disease course and/or modified by the treatment.

The investigators believe that understanding these neutrophil perturbations can lead to better monitoring of disease activity. Ultimately, the investigators may propose more targeted anti-inflammatory therapies which would be better tolerated by patients. the investigators also can identify new markers for disease activity which allow clinicians to define a better therapeutic strategy.

DETAILED DESCRIPTION:
A - Specific Aims General aim: This project is designed to study physiopathological mechanisms involved in GPA at the cellular and molecular level. the investigators want to study neutrophils as prognostic factors and determine the implication of PR3, the major autoantigen in the resolution phase of inflammation.

the investigators' working hypothesis is that structural and functional analysis of PR3 in neutrophils will help the investigators to unravel its role in GPA. Hence, our long-term objective is to better understand the mechanisms involved in the modulation of PR3 expression at the membrane of neutrophils in order to inhibit their activation and propose novel anti-inflammatory therapeutic strategies adapted to GPA.

Present project: The investigators recently demonstrated that in human neutrophils i) PR3 can be expressed at the membrane of neutrophils during apoptosis in the absence of degranulation, ii) PR3 is a member of a molecular scaffold comprising phospholipidscramblase1 (scramblase) and calreticulin externalized during apoptosis, iii) apoptosis-induced PR3 membrane expression impairs macrophage reprogramming after phagocytosis of apoptotic neutrophils The investigators' hypothesis is that PR3 might have specific molecular partners which can facilitate its externalization and/or its persistence at the plasma membrane during neutrophil apoptosis thus potentiating its auto-antigenic capacity.

The specific aims are:

1. Characterization of apoptosis in neutrophils from GPA patients
2. Analysis of PR3 partners (CD16, CD11b, Calreticulin, Phospholipidscramblase1) or co-expressed protein of interest in inflammation (AnnexinA1,) expression in neutrophils from patients with GPA compared to healthy controls
3. Identification of new partners of PR3 in neutrophils
4. Analysis of the proteome of neutrophils from GPA patients

B. Background and Significance 1.1. Introduction GPA is a systemic vasculitis which is mainly associated with anti-PR3 ANCA. The role of activated neutrophils in vasculitis lesions is suggested by their presence in perivascular infiltrates, especially in kidney glomeruli and in the lung.

PR3 is a serine protease first described within azurophilic granules of neutrophils which are NOT supposed to fuse with the plasma membrane but are released within the phagolysosome after phagocytosis of the pathogen. We have shown for the first time that the subcellular localization of PR3 was not restricted to azurophilic granules, as previously thought, but that PR3 was localized in secretory vesicles, a highly mobilizable compartment, thus explaining the presence of PR3 at the surface of resting isolated neutrophils. Moreover, a high percentage of neutrophils expressing PR3 observed in vasculitis patients could be considered as a risk factor for vasculitis. This high expression of membrane PR3 in patients with GPA resulted in an increase in ANCA-induced respiratory burst in neutrophils thus enhancing the inflammatory process. In vitro the binding of ANCA to PR3 trigger the respiratory burst, degranulation and the release of pro-inflammatory cytokines.

Because PR3 membrane expression is an important pathophysiological event in GPA since it is a prerequisite for the subsequent activation of neutrophils by ANCA, we sought to determine mechanisms involved in PR3 membrane expression. In neutrophils, we demonstrated that apoptosis triggered a significantly increased membrane PR3 expression without degranulation. In these experiments, we failed to detect MPO at the membrane of neutrophils. Our results differ from previously reported data showing that both MPO and PR3 were externalized during apoptosis because of the translocation of azurophilic granules to the plasma membrane. This phenomenon seems to occur when neutrophils undergo late apoptosis and secondary necrosis, leading to expression of all granule proteins on the cell surface.

Apoptosis-induced PR3 externalization could be of great relevance in the pathophysiology of GPA because PR3, which was supposed to be an intracellular antigen, is thus exposed at the plasma membrane of apoptotic cells thus amplifying its pro-inflammatory potential, its immunogenic properties and interfering with macrophage phagocytosis. We have also demonstrated that during apoptosis PR3 expression is associated with the expression of calreticulin, a well-known "eat-me signal". We have finally evidenced that the presence of PR3 impairs the reprogramming of macrophage to an anti-inflammatory profile after phagocytosis of apoptotic cells through the CRT/LRP pathway.

It can be hypothesized that the expression of the complex PR3/scramblase/CRT and other partners (CD11b, CD16) at the surface of apoptotic neutrophils could constitute good prognosis markers.. Gene array studies have pointed out a deregulation of neutrophils in GPA. We make the hypothesis that the proteome of neutrophils of GPA patients would be very informative of its activation state, survival state and that it could be a biological marker of clinical severity.

It is thus pertinent to study the deregulation of neutrophils during their all life cycle: their oxidative burst under activation, their physiologic apoptosis, the expression of PR3 partners. This study will be performed in neutrophils from patients with GPA compared to age and sex adjusted healthy controls.

C. Preliminary studies Analysis of apoptosis in neutrophils from GPA patients In the literature, neutrophils from patients with ANCA associated vasculitis (AAV) were found to have a disturbed TNFα-induced apoptosis and tends to have a higher rate of apoptosis than controls. However, published data on physiologic apoptosis which is the spontaneous apoptosis that neutrophils undergo in the absence of exogenous stimuli is contradictory. When calf foetal serum is added in medium, neutrophils from GPA patients display a similar apoptosis rate than controls. When the serum of patients is used, neutrophils from AAV patients in remission have a higher survival rate in vivo than controls, and this difference disappear when normal serum is used. These results are in agreement with the discovery that GPA patients have a high expression of PCNA which is associated with survival. Therefore, we want to study the apoptosis rate of neutrophils in GPA at diagnosis, during relapse and after remission on whole blood. These results will be compared to age and sex matched controls. Apoptosis will be evaluated by the phosphatidylserine externalization measured by flow cytometry after annexin-V labelling and 7-AAD staining on CD15+ cells. PCNA expression will be also investigated at the different clinical stage and proteomic profile of apoptotic neutrophils will be performed.

Analysis of scramblase/ Calreticulin expression in neutrophils from GPA patients In a cellular model (RBL cell line), we have demonstrated that scramblase extinction by shRNA was associated with a decreased expression of phosphatidylserine during apoptosis and that PR3 apoptosis induced expression was also impaired (unpublished data). We were also able to demonstrate that in vitro scramblase and PR3 physically interact. During apoptosis, PR3 is also associated with calreticulin at the membrane of neutrophils. These data suggest that the association PR3/Scramblase/Calreticulin form a molecular scaffold which is a functional platform which could interfere with recognition pathways (like CRT/LRP) between macrophages and apoptotic neutrophils. The expression of these partners at the neutrophil membrane during apoptosis will be investigated in patients at diagnosis and when remission is obtained.

Research design and Methods:

1. Characterization of apoptosis in neutrophils from GPA patients We will determine apoptosis rate of neutrophils in whole blood.

   Methodology:

   Research will be performed both on neutrophils isolated from healthy control donors obtained in the French Blood Institute (Etablissement Français du Sang) and from vasculitis patients from the Department of Internal Medicine of Cochin Hospital headed by Professor Loïc Guillevin.

   Apoptosis will be induced "physiologicaly" in whole blood by overnight incubation at 37°C.

   Phosphatidylserine externalization will be measured by flow cytometry after annexin-V labeling associated with 7-AAD staining for CD15+ cells.

   Western blot analysis using a specific antibody against PCNA will also be used to visualize its expression.
2. Analysis of scramblase, PR3, calreticulin, AnnexinA1, expression in apoptotic neutrophils from GPA patients We will determine the membrane expression of PR3, CRT, PLSCR, AxA1, in apoptotic neutrophils in the different subsets of neutrophils: non apoptotic ones (AnnexinV-, 7AAD-), early apoptotic neutrophils (AnnexinV+, 7AAD-) and late apoptotic neutrophils (AnnexinV+, 7AAD+). This determination will be done for patients at the time of diagnosis (in active state; BVAS>3) and at remission.

   Methodology
   * Neutrophils will be isolated from blood using Dextran gradient and Ficoll.
   * Investigation of PR3, CRT, PLSCR, AxA1, membrane expression will be measured on isolated neutrophils by flow cytometry after overnight incubation at 37°C with assessment of apoptosis by annexin-V labeling and 7AAD staining.
3. Study of the respiratory burst in neutrophils of GPA patients One of the main functions of neutrophils is the production of reactive oxygen species, we will determine the oxidative metabolism of neutrophils due to different stimuli (f-MLP, opsonized zymosan beads by complement, opsonized zymosan beads by IgG, PMA) with or without a previous priming by TNFα.

   Methodology:

   Exploration of the respiratory burst will be done in whole blood with a chemoluminescent (luminol) technique. Neutrophils will be primed by TNFα or stimulated without priming. The burst response will be analysed during 90 minutes after stimulation.
4. Deregulation of neutrophil Cytokinome Neutrophils are capable to synthetize a large number of cytokines (IL-1, TNFα, IL-6, IL-12), growth factors like GM-CSF and chimiokines like IL-8. More recently it has been shown that neutrophils are also great producers of BAFF (B-cell activating factor) and that production is superior to those by monocytes or dendritic cells when stimulated by INF-γ. In GPA serum BAFF levels have been shown to be higher than controls and recently targeting B-lymphocytes therapeutics have confirmed in large controlled trials their importance in AAV.

   Methodology:

   Serum of patients will be collected at the same time than neutrophils. They will be analyzed using BD™ Cytometric Bead Array (CBA) with detection of IL-8, IL-1β, IL-6, IL-10, TNF, and IL-12p70. Neutrophils which will be isolated as in 1) will be stimulated by INF-γ, LPS and G-CSF to analyze their production and secretion of BAFF/BlyS determined by ELISA.
5. Deregulation of neutrophil Proteome and functional study of new PR3 partners Gene array studies have shown a probable deregulation of neutrophils in AAV, in this study we will study this deregulation at the protein level.

Methodology:

To study the proteome of GPA patient when active and in remission compared to healthy controls we will use a differential in gel electrophoresis of cytosolic samples of neutrophils obtained by sonication. Identification of proteins of interest will be done by mass spectrometry MALDI-TOF-TOF. Functional validation of these proteins by over-expression or siRNA extinction will be performed.

ELIGIBILITY:
Inclusion Criteria:

For patients with GPA

* Systemic or localized GPA with ACR (American College of Rheumatology) criteria.
* BVAS > 3.
* ANCA anti-PR3 or anti-MPO
* Consent form signed

For patients with MPA

* Systemic MPA with Chapel Hill criteria.
* BVAS > 3.
* ANCA anti-MPO
* Consent form signed

For patients with EGPA

* Systemic EGPA with ACR (American College of Rheumatology) criteria.
* BVAS > 3.
* ANCA anti-PR3 or anti-MPO
* Consent form signed

For atherosclerotic patients

* Ischemic stroke
* Coronary heart attack
* Peripheral vascular disease responsible for intermittent claudication
* Carotid Stenosis

Exclusion Criteria:

* Pregnancy
* <18 yr
* Malignancy
* Infectious diseases: HIV, HBV, HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: GPA (Granulomatosis with polyangiitis) patients and MPA ( Microscopic Polyangiitis) with an active disease at inclusion
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2012-05-25 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
level of neutrophils | At Day 0
  Proteomic analysis of neutrophils compared to healthy donors and MPA (microscopic polyangiitis) patients

CONTACTS AND LOCATIONS:
Locations (1):
- Cochin Hospital, Paris, France

REFERENCES:
- [Background] Millet A, Martin KR, Bonnefoy F, Saas P, Mocek J, Alkan M, Terrier B, Kerstein A, Tamassia N, Satyanarayanan SK, Ariel A, Ribeil JA, Guillevin L, Cassatella MA, Mueller A, Thieblemont N, Lamprecht P, Mouthon L, Perruche S, Witko-Sarsat V. Proteinase 3 on apoptotic cells disrupts immune silencing in autoimmune vasculitis. J Clin Invest. 2015 Nov 2;125(11):4107-21. doi: 10.1172/JCI78182. Epub 2015 Oct 5. PMID 26436651
- [Derived] Amsler J, Everts-Graber J, Martin KR, Roccabianca A, Lopes C, Tourneur L, Mocek J, Karras A, Naccache JM, Bonnotte B, Samson M, Hanslik T, Puechal X, Terrier B, Guillevin L, Neel A, Mouthon L, Witko-Sarsat V. Dysregulation of neutrophil oxidant production and interleukin-1-related cytokines in granulomatosis with polyangiitis. Rheumatology (Oxford). 2024 Aug 1;63(8):2249-2258. doi: 10.1093/rheumatology/kead578. PMID 37947315